CLINICAL TRIAL: NCT05009134
Title: Influences of Allergic Rhinitis and Allergen Immunotherapy on Human Antibody Responses to SARS-CoV-2 Vaccination
Brief Title: Influences of Allergic Rhinitis and Allergen Immunotherapy on SARS-CoV-2 Vaccination
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Zheng Liu, Professor of Otolaryngology-Head & Neck Surgery, Deputy Dean of Tongji Hospital, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Huazhong University of Science and Technology
Other Study IDs: ENT-ALLERGY-01
Record Dates: First submitted 2021-08-10; First posted 2021-08-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Allergic Rhinitis; Allergen Immunotherapy; SARS-CoV-2
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples will be collected at baseline (prior to vaccinate), 7 and 30 after first vaccine, and, 7 and 30 after second vaccine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: 18-55 years, healthy
  Interventions: Biological: There is no intervention in this study.
- Allergic rhinitis: patients with AR without AIT
  Interventions: Biological: There is no intervention in this study.
- Allergen immunotherapy: patients with AR with AIT for more than 1 year
  Interventions: Biological: There is no intervention in this study.

INTERVENTIONS:
Biological: There is no intervention in this study. — There is no intervention in this study.

SUMMARY:
The study is designed to assess whether allergic rhinitis and allergen immunotherapy affect the humoral response to SARS-CoV-2 Vaccination in adults. This is a prospective study enrolling a total of approximately 120 subjects, 18-55 years old.

DETAILED DESCRIPTION:
Background: Allergic rhinitis (AR) is a disorder caused by hypersensitivity of the immune system to harmless allergens in the environment, which represents a global public health problem affecting up to 20-50% of the population. Allergen immunotherapy (AIT) is the only effective treatment that not only has disease-modifying property but also confers long-term clinical benefit after cessation of treatment for AR patients. Vaccination is one of the most powerful interventions for reducing disability and death caused by infectious disease. Immunization with the inactivated SARS-CoV-2 Vaccine remains the most effective strategy to combat COVID-19 infections. Nevertheless, the influences of allergic rhinitis and allergen immunotherapy on SARS-CoV-2 vaccination are still unknown.

Objectives: To investigate if AR and AIT will influence the humoral response to SARS-CoV-2 vaccination in adults.

Design and trial size: This is a prospective study. A total of approximately 120 subjects, 18-55 years old, including 40 healthy subjects, 40 patients with AR without AIT, and 40 patients with AR with AIT for more than 1 year, will be enrolled in this study.

Intervention and duration: All of the study participants will be vaccinated with an 2 doses inactivated vaccine against SARS-CoV-2 (COVILO). Peripheral blood samples will be collected at baseline (prior to vaccinate), 7 and 30 after first vaccine, and, 7 and 30 after second vaccine. One-month additional data analysis leads to the trial duration of 3 months.

ELIGIBILITY:
Inclusion Criteria:

18-55 years; healthy subjects, patients with AR without AIT, or patients with AR with AIT for more than 1 year

Exclusion Criteria:

1. who infected with COVID-19 previously
2. Cannot finish the follow up
3. Previous allergic to other vaccines
4. who have had severe immunologic, cardiac, liver or metabolic disease, tumors, allergic diseases, or chronic infection,
5. pregnancy or breastfeeding
6. Suffered from airway infection or severe infectious diseases in the past 3 months, prior to this study.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: 18-55 years; healthy subjects, patients with AR without AIT, or patients with AR with AIT for more than 1 year
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2022-03-20 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Virus-specific antibodies levels in serum and humoral immune response as measured by ELISA or HAI assay | Jun 2021-Aug 2021
  Virus-specific antibodies levels in serum and humoral immune response as measured by ELISA or HAI assay
Frequencies and numbers of circulating T cell subsets, B cell subsets, dendritic cells, NK cells in peripheral blood | Jun 2021-Aug 2021
  Frequencies and numbers of circulating T cell subsets, B cell subsets, dendritic cells, NK cells in peripheral blood
Levels of antigen-specific IgE and IgG4, IFN-γ, IL-4, IL-5, IL-10, IL-17A, and IL-21 in serum detected by ELISA | Jun 2021-Aug 2021
  Levels of antigen-specific IgE and IgG4, IFN-γ, IL-4, IL-5, IL-10, IL-17A, and IL-21 in serum detected by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Liu, Doctor, Study Chair — Tongji Hospital
Locations (1):
- Department of ENT, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao X, Luo K, Wang D, Wei Y, Yao Y, Deng J, Yang Y, Zeng Q, Dong X, Xiong L, Gong D, Lin L, Pohl K, Liu S, Liu Y, Liu L, Nguyen THO, Allen LF, Kedzierska K, Jin Y, Du MR, Chen W, Lu L, Shen N, Liu Z, Cockburn IA, Luo W, Yu D. T follicular helper 17 (Tfh17) cells are superior for immunological memory maintenance. Elife. 2023 Jan 19;12:e82217. doi: 10.7554/eLife.82217. PMID 36655976
- [Derived] Yao Y, Huang A, Deng YK, Liu Y, Zhu HY, Wang N, Wang ZZ, Zhu RF, Yu D, Liu Z. Allergen Immunotherapy Reverses Immune Response to SARS-CoV-2 Vaccine in Patients with Allergic Rhinitis: A Prospective Observational Trial. Am J Respir Crit Care Med. 2022 Sep 15;206(6):780-783. doi: 10.1164/rccm.202203-0608LE. No abstract available. PMID 35649178